CLINICAL TRIAL: NCT03814070
Title: Prosthesis and Implant Survival in Immediately Loaded Full Arch Restorations Using Fiber Reinforced Versus Non-reinforced Temporary Frameworks: A Randomized Clinical Trial
Brief Title: Prosthesis and Implant Survival in Immediately Loaded Temporary Full Arch Restorations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nermeen Ahmed Hassan (Other)
Responsible Party: Sponsor-Investigator, Nermeen Ahmed Hassan, PhD candidate, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nermeen Ahmed Hassan
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Completely Edentulous Patients

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-reinforced full arch acrylic restorations (Active Comparator)
  Interventions: Procedure: No framework
- full arch acrylic restorations with fiber-reinforced framework (Experimental)
  Interventions: Procedure: Fiber-reinforced framework

INTERVENTIONS:
Procedure: Fiber-reinforced framework — Glass fiber- reinforced framework is to be picked up over the implant abutments to strengthen the full arch acrylic restorations
  Arms: full arch acrylic restorations with fiber-reinforced framework
Procedure: No framework — Non-reinforced acrylic full arch prosthesis is to be picked up directly over the implant abutments.
  Arms: Non-reinforced full arch acrylic restorations

SUMMARY:
In immediate loading of implants of completely edentulous patients, the most common post-surgical complication following the surgery noted in the dental literature is fracture of the provisional restoration with rates ranging from 4.17% to 41%. Most of these fractures occur because polymethyl methacrylate (PMMA) materials are inadequate and have low rigidity to withstand extended periods of heavy occlusal use.

Fractures of full arch provisional restorations during healing are concerning, because they eliminate cross-arch stabilization and disrupt stress distribution patterns which might jeopardize implant osseointegration affecting the survival rates for implants. Therefore, it is important to look for another material that has higher rigidity than PMMA and can withstand masticatory forces for extended periods without fractures or load concentration on the implants during the osseointegration period.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous patients.
* Patients with proper amount of attached gingiva (≥2 mm)

Exclusion Criteria:

* Patients having a medical condition that absolutely contraindicates implant placement.
* Patients with uncontrolled diabetes, assessed by measuring glycosylated hemoglobin (HbA1c). (greater than 6.4 percent)
* Potentially uncooperative patients who are not willing to go through the proposed interventions.
* Moderate-to-heavy daily smokers* (who report consuming at least 11 cigarettes/day).
* Patients with history of bruxism
* If insertion torque for the implants is less than 35 Ncm

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Prosthesis survival | 4 months
  Clinical evaluation of any fracture in the prosthesis

SECONDARY OUTCOMES:
Implant survival | 4 months
  Clinical evaluation of implant loss
Peri-implant crestal bone loss during healing | 4 months
  Crestal bone loss around implants is to be measured using periapical x ray with parallel technique in millemeters